CLINICAL TRIAL: NCT04920643
Title: High-exchange ULTrafiltration to Enhance Recovery After Pediatric Cardiac Surgery (ULTRA): A Canadian Randomized Controlled Trial
Brief Title: High-exchange ULTrafiltration to Enhance Recovery After Pediatric Cardiac Surgery
Acronym: ULTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Dr. David Horne, Congenital Cardiac Surgeon, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IWKHealthC
Record Dates: First submitted 2021-05-30; First posted 2021-06-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Ultrafiltration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Exchange Ultrafiltration (Experimental): Subzero-Balance Simple Modified Ultrafiltration (60ml/kg/hour)
  Interventions: Procedure: Ultrafiltration
- Low-Exchange Ultrafiltration (Active Comparator): Subzero-Balance Simple Modified Ultrafiltration (6ml/kg/hour)
  Interventions: Procedure: Ultrafiltration

INTERVENTIONS:
Procedure: Ultrafiltration — Ultrafiltration is used during cardiac surgery with cardiopulmonary bypass to remove both fluid and small molecules such as inflammatory cytokines from the patient's circulation.

SUMMARY:
Malformations of the heart are common; 1.35 million infants are born each year with congenital heart disease. Many of these defects carry a considerable threat to the individual's quality of life as well as survival. Along with focused medical management, surgical repair remains a standard of care for more than 25,000 infants and children each year in the United States and Canada. The care of individuals with congenital heart disease is highly complex and has significant risks of morbidity and mortality. Most cardiac operations require the use of cardiopulmonary bypass (CPB, also known as the heart-lung machine) to safely access the inner chambers of the heart. CPB itself has been well documented to cause significant inflammation and hemodilution as the individual's blood is passed through a foreign circuit. This inflammatory response can lead to fluid overload, distributive shock and potential end-organ dysfunction in the heart, lungs, kidneys, brain, liver or bowels. These organ dysfunctions may culminate in post-operative low cardiac output syndrome (LCOS), prolonged ventilation time, prolonged intensive care unit (ICU) stay and can contribute to mortality.

Dampening the inflammatory response from CPB has been a focus of research interest for years. Intra-operative ultrafiltration has been used to remove excess fluids and filter off inflammatory cytokines during cardiac operations. Over 90% of children's heart centers in the world utilize some form of ultrafiltration (mostly some form of modified ultrafiltration), but there are wide variations in published ultrafiltration protocols (none of which are combination SBUF-SMUF in children). Ultimately, this project seeks to provide high-quality evidence that the immunologic and clinical effects of combination SBUF-SMUF are rate dependent. Therefore, a randomized study directly comparing a high-exchange SBUF-SMUF (60ml/kg/hr) and a low-exchange SBUF-SMUF (6ml/kg/hr) can identify which is the optimal ultrafiltration protocol to enhance post-operative clinical outcomes for this patient population. The expected data and results could be immediately applicable to improve recovery after heart surgery for infants and children across Canada and the rest of the world at large.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart patients (2.5 - 15kg) have consented for a planned cardiac surgery procedure requiring cardiopulmonary bypass.
* Parent or legal substitute decision-maker informed written consent to participate in the study.

Exclusion Criteria:

* Patient or family refusal to participate.
* Patient over 15kg (Fontan or Glenn patients will be considered up to 18kg)
* No planned use of cardiopulmonary bypass
* Isolated ASD repair
* Known severe hematologic abnormality such as sick cell anemia, thalassemia, haemophilia A or B, von Willebrand disease or other.
* Known genetic syndrome with severe neurologic or multi-organ abnormalities and immune dysfunction such as DiGeorge Syndrome, Trisomy 18 or 13, Noonan syndrome. (Trisomy 21 may be included in the study).
* Known immunodeficiency syndrome or bone marrow pathology.
* Severe liver or renal disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Peak Vasoactive-Ventilation Renal Score | Up to 5 days

SECONDARY OUTCOMES:
Vasoactive Inotrope Score | Up to 5 days
  Taken in time series at ICU admission, 0, 12, 24, 36, 48, 72, 96 and 120 hours.
Ventilation Index | Up to 5 days
  Taken in time series at ICU admission, 0, 12, 24, 36, 48, 72, 96 and 120 hours.
Oxygenation Index | Up to 5 days
  Taken in time series at ICU admission, 0, 12, 24, 36, 48, 72, 96 and 120 hours.
Ventilation Time | Up to 28 days
Ventilator Free Days | Up to 28 days
Low Cardiac Output Syndrome | Up to 3 days
  Defined by any one of the following within the first 72 post-operative hours:
  * Lactate > 4mM with oxygen extraction >35% (SaO2 - ScvO2/ SaO2)
  * VIS > 15.0 with oxygen extraction >35% (SaO2 - ScvO2/ SaO2)
  * Mechanical circulatory support requirement
Vasoplegic Shock | Up to 3 days
  Defined by any one of the following with the first 72 post-operative hours:
  * Lactate > 4mM with oxygen extraction <25% (SaO2 - ScvO2/ SaO2)
  * VIS > 15.0 with oxygen extraction <25% (SaO2 - ScvO2/ SaO2)
Inotrope Dependence | Up to 2 days
  Vasoactive-inotrope score at 48 hours equal to or greater than that at ICU admission.
Inotrope Free Days | Up to 28 days
C-Reactive Protein Concentrations | Measured at 1 day
Composite Outcome of mechanical circulatory support, acute renal failure, prolonged intubation and operative mortality. | Up to 30 days
Cytokine Concentration (Patient Plasma) | Up to 1 day
  C3, C3a, C3b, C5, C5a, IL-1, IL1-Ra, IL-6, IL-10, TNF, CXCL-8 among others. The final selection of mediators will be subject to final pilot study results and assay availability. Taken at baseline, 0 hours and 24 hours after CPB.
Loop Diuretic Use | Up to 7 days
  Total loop diuretic (mg/kg), measured in furosemide equivalents, during the first 7 post-operative days.
Peak Vasoactive-Inotrope Score | Up to 5 days
Peak Ventilation Index | Up to 5 days
Peak Oxygenation Index | Up to 5 days
Prolonged Intubation | Up to 28 days
  Mechanical ventilation for more than 7 days
Inotrope Time | Up to 28 days
Acute Kidney Injury | Up to 28 days
  KDIGO Criteria
ICU Length of Stay | Up to 30 days
Hospital Length of Stay | Up to 60 days
Haptoglobin (Plasma) | Up to 1 day
Complete blood count | Up to 5 days
Lactate | Up to 5 days
  Measured by arterial blood gas (mM)
Creatinine | Up to 5 days
  Blood Concentration (uM)
Vasoactive-Ventilation Renal Score | Up to 5 days
  Taken in time series at ICU admission, 12, 24, 36, 48, 72, 96 and 120 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bierer J, Stanzel R, Henderson M, Sett S, Horne D. Ultrafiltration in Pediatric Cardiac Surgery Review. World J Pediatr Congenit Heart Surg. 2019 Nov;10(6):778-788. doi: 10.1177/2150135119870176. PMID 31701831
- [Derived] Bierer J, Stanzel R, Henderson M, Krmpotic K, Andreou P, Marshall JS, Sapp J, Horne D. High-exchange ULTrafiltration to enhance recovery after paediatric cardiac surgery (ULTRA): study protocol for a Canadian double-blinded randomised controlled trial. BMJ Open. 2024 Aug 28;14(8):e080597. doi: 10.1136/bmjopen-2023-080597. PMID 39209495